CLINICAL TRIAL: NCT03385161
Title: Intraprostatic Injection of Botulinum Toxin A Versus Ethanol for Treatment of Patients With Benign Prostatic Hyperplasia Refractory to Medical Treatment
Brief Title: Intraprostatic Injection of Botulinum Toxin A Versus Ethanol for Treatment of Patients With Benign Prostatic Hyperplasia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Mohammed Said ElSheemy, Associate Professor of Urology, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 61352
Record Dates: First submitted 2017-12-20; First posted 2017-12-28 (Actual); Last update posted 2017-12-28 (Actual); Status verified 2017-12

CONDITIONS: Male; Ultrasonography; Botulinum Toxins, Type A; Injection; Complications, Infection; Prostatic Hyperplasia
Keywords: ethanol ablation of the prostate; Benign prostatic hyperplasia (BPH); Prostate; Ethanol; Transrectal; BPH; onaBoNT-A; Botox; Lower urinary tract symptoms; Botulinum toxin; OnabotulinumtoxinA; Quality of life; IPSS; Randomised controlled study
MeSH Terms: conditions — Infections; Prostatic Hyperplasia; Lower Urinary Tract Symptoms | interventions — Botulinum Toxins, Type A; onabotulinum toxin A; Ethanol

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: Only the surgeon during injection knows the active material
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- botulinum toxin A (Active Comparator): Intraprostatic injection of botulinum toxin A (onabotulinumtoxinA; 100 IU) through transrectal ultrasonography.
  One vial (100 IU) is dissolved in 10 ml saline and injected in the transition zone of each lobe of the prostate in 3 sites; basal, middle and apical.
  one gm intramuscular ceftriaxone started and continued 3 days. A rectal enema performed the night before the procedure. The anal area sterilized A 21 gauge needle was introduced to the prostate.
  Interventions: Procedure: Botulinum toxin A
- Ethanol (Active Comparator): Intraprostatic injection of dehydrated ethanol through transrectal ultrasonography.
  An amount equal to 25% of prostate volume was injected distributed over 6-8 sites among both prostatic lobes with an average of 2 ml per site.
  one gm intramuscular ceftriaxone started and continued 3 days. A rectal enema performed the night before the procedure. The anal area sterilized A 21 gauge needle introduced to the prostate.
  Interventions: Procedure: Ethanol

INTERVENTIONS:
Procedure: Botulinum toxin A
  Other Names: onaBONT/A; botox; onabotulinumtoxinA
  Arms: botulinum toxin A
Procedure: Ethanol
  Other Names: dehydrated ethanol
  Arms: Ethanol

SUMMARY:
To compare safely and efficacy of intraprostatic injection of botulinum toxin A versus ethanol for treatment of benign prostatic hyperplasia (BPH).

DETAILED DESCRIPTION:
To compare safely and efficacy of transrectal intraprostatic injection of botulinum toxin A versus ethanol for treatment of symptomatic benign prostatic hyperplasia (BPH) refractory to medical treatment.

ELIGIBILITY:
Inclusion Criteria:

* international prostate symptoms score (IPSS) > 7
* Qmax < 15
* Patients with refractory symptomatic BPH to medications
* patients high risk for surgery or unwilling to do surgery

Exclusion Criteria:

* bladder stones
* acute or chronic urinary retention
* urethral stricture
* bladder or prostatic carcinoma.
* Neurogenic bladder dysfunctions

Ages: 50 Years to 75 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Prostate is only in males
Enrollment: 90 (Actual)
Dates: Start 2013-12 (Actual); Primary Completion 2015-06 (Actual); Study Completion 2017-06 (Actual)

PRIMARY OUTCOMES:
International prostate symptom score (IPSS) | 1, 3, 6 months and one year
  7 items Questionnaire with a score range from 0 - 35 (5 points for each item) A score of 35 is considered the worst The score is calculated during each period of follow-up The difference in the score in each group will be compared versus each other to detect any significant difference between both groups

SECONDARY OUTCOMES:
Maximum flow rate (Qmax) | 1, 3, 6 months and one year
  The peak flow rate measured during flowmetry (mL/Sec) Increase in the flow rate is considered improvement The Qmax is calculated during each period of follow-up by flowmetry The difference in the Qmax in each group will be compared versus each other to detect any significant difference between both groups
Prostate volume | 1, 3, 6 months and one year
  Prostate volume (PV) will be measured by transrectal US (Cubic cm) Decrease in size is considered improvement The PV is calculated during each period of follow-up The difference in the PV in each group will be compared versus each other to detect any significant difference between both groups
quality of life (QoL) | 1, 3, 6 months and one year
  one items Questionnaire It is the QoL portion of the International prostate symptom score (IPSS) The score range from 0 - 6 A score of 6 is considered the worst The score is calculated during each period of follow-up The difference in the score in each group will be compared versus each other to detect any significant difference between both groups

OTHER OUTCOMES:
retention of urine | 1, 3, 6 months and one year
  Significant difference between the rate (%) of development of retention of urine in both groups during follow-up
Other lines of treatment including TURP | 1, 3, 6 months and one year
  Significant difference between the rate (%) of required TURP and other lines of treatment in both groups (due to failure of studied intervention to improve symptoms of the patient )

CONTACTS AND LOCATIONS:
Overall Officials: Mohammed S ElSheemy, Ass. Prof., Principal Investigator — Cairo University
Locations (1):
- Cairo University Hospitals, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Totaro A, Pinto F, Pugliese D, Vittori M, Racioppi M, Foschi N, Bassi PF, Sacco E. Intraprostatic botulinum toxin type "A" injection in patients with benign prostatic hyperplasia and unsatisfactory response to medical therapy: A randomized, double-blind, controlled trial using urodynamic evaluation. Neurourol Urodyn. 2018 Mar;37(3):1031-1038. doi: 10.1002/nau.23390. Epub 2017 Aug 25. PMID 28840969
- [Result] Marberger M, Chartier-Kastler E, Egerdie B, Lee KS, Grosse J, Bugarin D, Zhou J, Patel A, Haag-Molkenteller C. A randomized double-blind placebo-controlled phase 2 dose-ranging study of onabotulinumtoxinA in men with benign prostatic hyperplasia. Eur Urol. 2013 Mar;63(3):496-503. doi: 10.1016/j.eururo.2012.10.005. Epub 2012 Oct 12. PMID 23098762
- [Result] Magno C, Mucciardi G, Gali A, Anastasi G, Inferrera A, Morgia G. Transurethral ethanol ablation of the prostate (TEAP): an effective minimally invasive treatment alternative to traditional surgery for symptomatic benign prostatic hyperplasia (BPH) in high-risk comorbidity patients. Int Urol Nephrol. 2008;40(4):941-6. doi: 10.1007/s11255-008-9394-z. Epub 2008 May 14. PMID 18478352
- [Result] Sakr M, Eid A, Shoukry M, Fayed A. Transurethral ethanol injection therapy of benign prostatic hyperplasia: four-year follow-up. Int J Urol. 2009 Feb;16(2):196-201. doi: 10.1111/j.1442-2042.2008.02205.x. Epub 2008 Nov 27. PMID 19054163